CLINICAL TRIAL: NCT02067052
Title: New Strategy for the Treatment of Vulvar Cancer Employing Sentinel Scintigraphy, Surgery, Chemotherapy, and Radiotherapy
Brief Title: New Strategy for the Treatment of Vulvar Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NP 245/12
Record Dates: First submitted 2013-08-30; First posted 2014-02-20 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Vulvar Neoplasm
Keywords: Vulvar neoplasm; sentinel nodes; chemotherapy; radiotherapy
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Surgical Procedures, Operative; Radiotherapy; Drug Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Advanced vulvar cancer: Patients with advanced-stage tumors.
  Interventions: Procedure: Surgery, radiotherapy and chemotherapy
- Early-stage vulvar cancer: Patients with early-stage tumors
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery, radiotherapy and chemotherapy — Surgery: vulvectomy and lymphadenectomy Radiotherapy: 180 cGy / day per 5 days untill maximum dose 4500 - 5940 cGy Chemotherapy: vulvectomy, lymphadenectomy
  Groups: Advanced vulvar cancer
Procedure: Surgery — Vulvectomy & lymphadenectomy
  Groups: Early-stage vulvar cancer

SUMMARY:
Vulvar cancer is a rare disease that is treated with surgery, radiation and chemotherapy. When tumors are large (greater than 4 cm) or compromise the urethra (urine canal) and the anus, or when it is in the groin lymph nodes, surgery alone is not always able to be performed. In this circumstance, is necessary to add radiotherapy, chemotherapy or both .

So far it is not known the best sequence of treatment: surgery, chemotherapy or radiotherapy. The radical surgeries usually need long recovery term both in the region of the vulva and in the region of the groin lymph nodes. When it is performed, convalescence can delay other treatments, like radiotherapy and chemotherapy. On the other hand, the use of radiotherapy and chemotherapy as a first step treatment can result in a complete elimination of the disease in at least 30% of the cases or substantial reduction of its size, allowing less extensive surgery.

Investigators intend to use surgery, chemotherapy and radiotherapy in the treatment of vulvar cancer, but in a sequence that has not been studied, in order to increase benefits of these treatments, and reduce morbidity.

This study will be offered to patients who have disease of the vulva less than 4 cm (sentinel lymph node), or greater than 4 cm, or illness that compromises urethra and anus, or patients with disease in groin lymph nodes (glands).

1. On the eve of the surgery, investigators will inject dextran-70 labeled with technetium-99 m. Only patients with tumors smaller than 4 cm will do this procedure.
2. On the day of the surgery, the groin lymph nodes will be removed from the inguinal (groin) only. If lymph nodes are disease positive, the vulvectomy will not be performed at this time. Patients will be treated with radiation therapy with concomitant chemotherapy for approximately six weeks.
3. At the end of treatment with chemotherapy and radiotherapy, investigators will perform a surgery to remove the remaining tumor in the vulva.

DETAILED DESCRIPTION:
Vulvar cancer is a rare disease, striking 2 to 3/100,000 women annually. Dissemination of vulvar cancer is predominantly lymphatic; contiguous invasion also occurs, though much less frequently, whereas hematogenic dissemination is quite rare, especially in the absence of lymphatic spread. Approximately 25% - 35% of the patients in the early stages of the disease have metastasis. The standard treatment for the initial stages consists of radical excision of the vulvar tumor and uni- or bilateral inguinal-femoral lymphadenectomy. The latter procedure is necessary, for the non-removal of the lymph nodes, even if the disease seems undetectable in the nodes, may be fatal. Treatment effectiveness is good, and the likelihood of a recurrence of the disease in the inguinal-femoral lymph nodes is 1% - 10% . The determinants for prognosis are lymph node metastasis, tumor size and stage, depth of tumor invasion, and lymphovascular involvement. In locally advanced stages of the disease, involvement of the inguinal-femoral lymph node chain has consistently been demonstrated as the most important predictive factor of survival for the patient. In the last 30 years, changes in surgical treatment, such as separate incisions for the performance of inguinal-femoral lymphadenectomy and vulvectomy, preservation of the saphenous vein, and a more conservative excision of the primary vulvar lesion, have reduced morbidity. Despite of the advances in surgical treatment, postoperative complications are still paramount. The locally advanced disease generates greater morbidity when It involves the urethra, anus, or rectum, for wide resections, urinary derivations, or even pelvic exenteration is then required in order to obtain an adequate surgical margin. Such procedures entail not only mutilation of the patient but also a high morbidity rate. A concomitant chemotherapy and radiotherapy (CT-RT) regimen has been advocated for the patient with the purpose of downsizing the initial disease, thereby enabling a less mutilating complementary surgical treatment. A study by the Gynecologic Oncology Group used preoperative chemoradiation combined with cisplatin / 5-fluouracil for stage III and IV patients. After the treatment, only 2 (3%) out of 71 patients remained with a residual disease that showed no signs of shrinking. A study using data from 63 patients with advanced vulvar cancer (stages III and IV) who underwent either surgery (30 patients) first or CT-RT followed by surgery (33 patients), compared disease-free interval and survival and recurrence rates of the disease. The patients who received CT-RT treatment before surgery were younger and had larger vulvar growths and less lymph node metastasis. An important point is that the positive lymph node rate of the patients just prior to surgery was 83% for those initially treated with surgery and 54% for those treated with CT-RT plus surgery. This shows that, in advanced cases, CT-RT reduces the mass of positive lymph nodes, but the disease persists in more than 50% of the patients at the original site. Thus, excision of the lymph nodes is necessary to obtain as much control over the disease as possible. As the inguinal-femoral lymph node status is the most important prognostic factor in vulvar cancer, it is crucial to assess lymph node condition prior to therapy in order to select the best approach strategy for the disease. At present, the non-invasive techniques for the detection of lymph node metastasis are insufficiently accurate.The low accuracy of the non-invasive techniques for detecting inguinal-femoral lymph nodes, the importance of a diagnosis of lymph node metastasis in patients with vulvar cancer in the early stages, and lymphadenectomy morbidity open the way for the development of minimally invasive techniques, such as sentinel lymph node biopsy. Most advantages accruing from the adoption of sentinel lymph node biopsy are related to the lesser morbidity and mortality of the surgical procedure because of its reduced aggressiveness. Nevertheless, the desired information concerning the metastatic potential of the primary tumor is gained. In the case of other malignancies, such as breast cancer and melanoma, the sentinel lymph node false negative rate is low (0%-29%; 7.3% mean).A multicentric study that analyzed 403 patients with early-stage vulvar cancer (tumor up to 4 cm) showed that sentinel lymph node excision was a safe surgical procedure. A total of 259 patients with a negative sentinel lymph node were merely kept under observation after surgery. Recurrence in the inguinal region was 2.5% and the survival rate in a 3-year span was 97%. For the patients with a positive sentinel lymph node, a systematic inguinal-femoral lymph node excision was performed. These patients benefited from a high accuracy rate in the identification of micro-metastases with a predictive value close to 100%. A multicentric, observational study (GROINSS-V) subsequent to the study by Van der Zee et al. examined the evidence from 403 patients to determine the relationship between the metastasis size of the sentinel lymph node and the metastasis risk in non-sentinel lymph nodes and disease-free survival for early-stage vulvar cancer. It was impossible to establish a cutoff point below which the likelihood of a non-sentinel lymph node metastasis would be close to zero, thus insignificant. What was found, though, is that the larger the spread of the sentinel lymph node, the greater the probability of the other lymph nodes metastasizing. Besides, if the size of the sentinel lymph node was larger than 2 mm, the prognosis was bad. The present study has the main purpose of outlining a new strategy for vulvar cancer treatment, combining sentinel lymphoscintigraphy, chemotherapy, radiotherapy, and surgery in a way as yet untested. Objectives: Analysis of the complete pathological response in patients with an anatomicopathologic diagnosis of invasive vulva cancer, (stages II to IVa - FIGO), treated with surgery, chemiotherapy and radiotherapy in the following proposal: nodal debulking of the groin, chemoradiation and vulvectomy. Materials and methods: Patient enrollment: Twenty one consecutive patients from the Outpatient Clinic of Gynecological Oncology, Cancer Institute, São Paulo State (ICESP) with a diagnosis of vulvar carcinoma (early and advanced stages) will be studied as long as they agree to participate and sign an informed consent statement. All patients with tumors up to 4 cm in greatest diameter, uncompromised urethra or anus, and lymph nodes smaller than 15 mm in greatest diameter in scan images will be considered early-stage cases. Any other cases will be deemed advanced. In the first phase will be included 21 patients. If there are seven or more complete clinical and pathological response (patients who underwent surgical biopsy or surgical excision of the primary tumor site), the study continued with the inclusion of further 30 patients. Preoperative evaluation: Biopsy and anatomicopathologic, exam of the vulvar lesion, MRI of the pelvis and vulvar region. Clinical evaluation and surgical risk assessment: Patients with early-stage tumors: After sentinel lymph node analysis, patients with early-stage tumors will undergo systematic uni- or bilateral inguinal-femoral lymphadenectomy. In addition, an intraoperative frozen-section examination of the sentinel lymph node(s) will be conducted. On the eve of surgery, a peritumoral infusion will be made with dextran-70 marked with technetium-99 (a radiopharmaceutical from the Nuclear Medicine Service, Radiology Institute, School of Medicine, USP), volume of 0.1 ml per injection point (0.3 millicurie of technetium in each syringe) with total activity of 1.2 mCi in the 4 points. Following injection of the peritumoral infusion, the patients will undergo lymphoscintigraphy on the very same day in order to locate and record the inguinal lymph nodes marked by the radioactive substance. On the next day, patients will be injected with a patent blue infusion in the peritumoral area immediately before the inguinal-femoral lymphadenectomy. With the aid of a gamma-probe (endoprobe model 2002, France), the supposedly compromised lymph nodes will be removed first and then the others. Finally, the excision will be performed with a margin around the primary vulvar lesion. After its identification and excision, the sentinel lymph node will be dispatched for an intraoperative anatomicopathologic exam and classified as positive, negative, or suspicious for neoplastic cells. It will be handled immediately after excision, isolated, and subjected to transverse cuts at 1.5-mm-intervals. All fragments will be embedded in paraffin, cross-sectioned to obtain 3- µm-thick cuts, and stained with hematoxylin and eosin. if the initial sections of each and every paraffin block test negative, the lymph node will be additionally submitted to serial cuts at 50- µm-intervals up to the 6th level. From each interval of all of the fragments of all blocks, 2 sections will be taken, one to be stained with hematoxylin and eosin and the other to be mounted on a silane-coated slide, for immunohistochemical analysis. The initial sections of each block with the transverse cuts of the lymph node at 1.5-mm-intervals will be immunohistochemically examined for detection of cytokeratins anion exchanger 1 and 3(clone AE1/AE3, Dako). If the sentinel lymph nodes are disease-free, the surgical procedure continues with the resection of the vulvar lesion leaving a 1-cm-wide margin at the least (ideal margin=2 cm) and reaching into deeper planes. An intraoperative anatomicopathologic evaluation of the surgical margins is also carried out, and the patient will be excluded of the study. If the sentinel lymph nodes test positive, it is a case of advanced-stage tumor, and the surgery will be stopped at this time for further chemoradiation. Patients with advanced-stage tumors: Patients with advanced-stage tumors, the superficial fascia was incised, and all palpably enlarged nodes were removed and sent for frozen section. If proven positive for metastatic spread, no further groin dissection will be undertaken. If negative, a full inguina-femoral lymphadenectomy will be performed, and these patients will be excluded of the study. After nodal debulking of the groin, patients will receive cisplatin at 40 mg/m2 once a week for 7 weeks throughout radiotherapy, which will be performed at a 45-50-Gy dose, 1.8 Gy/day, 5 times a week. A dose reinforcement of over 5-10 Gy may be given depending on the number of compromised lymph nodes and the size or extracapsular extension of the lesion. The presence of obvious metastatic disease will require the inclusion not only of inguinal lymphatic drains but also of pelvic drains (even the iliac lymphatics) in the radiotherapy fields. If after reevaluation for surgery, the lesion shows no signs of shrinking, a dose reinforcement of up to 60 Gy or 66 Gy total dose will be administered. Surgery - resection of the vulvar lesion with a 1-cm-margin at least (ideal margin = 2 cm) including the deeper planes and evaluation of surgical margins by means of intraoperative anatomicopathologic exam - will be performed 30-120 days after the end of chemoradiotherapy. Data analysis: The following data will be analyzed: Perioperative data: % → Fisher's test; Immediate and late complications; Disease-free interval; Survival. Predicted duration of project:3 years

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological diagnosis of squamous cell carcinoma of the vulva;
* Performance status 0-3 (ECOG);
* Adequate bone marrow function, liver and kidney;

Exclusion Criteria:

- Patients with a history of treatment of other invasive cancers in the last 5 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty one consecutive patients with a diagnosis of vulvar carcinoma (early and advanced stages) will be studied.
  All patients with tumors up to 4 cm in greatest diameter, uncompromised urethra or anus, and lymph nodes smaller than 15 mm in greatest diameter in scan images will be considered early-stage cases. Any other cases will be deemed advanced.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Patological response | up to 24 months
  The groin lymph nodes will be removed from the inguinal (groin) only. If investigators find disease in the lymph nodes, the vulvectomy will not be performed at this time, but patients will be treated with radiation therapy with concomitant chemotherapy for a period of approximately six weeks.
  At the end of treatment with chemotherapy and radiotherapy, the investigators will perform a surgery to remove remaining tumour in the vulva followed by patological response evaluation.

SECONDARY OUTCOMES:
Inguinal lymphadenectomy-derived outcomes | up to 12 months
  Presence of active infection as defined by clinical determination of lymphocelle and wound breakdown

CONTACTS AND LOCATIONS:
Overall Officials: Altamiro R Dias Jr, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- USPauloGH, São Paulo, Brazil

REFERENCES:
- [Derived] Dias-Jr AR, Soares-Jr JM, de Faria MBS, Genta MLND, Carvalho JP, Baracat EC. Secondary healing strategy for difficult wound closure in invasive vulvar cancer: a pilot case-control study. Clinics (Sao Paulo). 2019;74:e1218. doi: 10.6061/clinics/2019/e1218. Epub 2019 Sep 2. PMID 31482981